CLINICAL TRIAL: NCT06080100
Title: RELIEF OF PSYCHOEMOTIONAL STRESS BEFORE REFRACTIVE LASER VISION CORRECTION SURGERY USING XENON SEDATION
Brief Title: RELIEF OF PSYCHOEMOTIONAL STRESS USING XENON SEDATION
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: The S.N. Fyodorov Eye Microsurgery State Institution (Other Government)
Responsible Party: Principal Investigator, Alexander Romanov, anesthesiologist, The S.N. Fyodorov Eye Microsurgery State Institution
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2023-10-01; First posted 2023-10-12 (Actual); Last update posted 2025-06-27 (Actual); Status verified 2025-06

CONDITIONS: Psychological Stress; Anesthesia; Anxiety; Xenon
Keywords: sedation; laser refractive interventions; anxiety; xenon
MeSH Terms: conditions — Stress, Psychological; Anxiety Disorders | interventions — Xenon

STUDY DESIGN:
Intervention Model Description: According to the latest data, the need for xenon analgosedation occurs in 10% of cases from all excimer laser operations. N= 1,96*10*90/25=70.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Main group (Active Comparator): patients with high anxiety and stress instability who underwent xenon analgosedation before refractive laser vision correction
  Interventions: Drug: Xenon
- Control group (Other): patients with high anxiety and stress instability who underwent local anesthesia using standard premedication with hydroxyzine (hydroxyzine) 25 mg.
  Interventions: Other: premedication hydroxyzine 25 mg

INTERVENTIONS:
Drug: Xenon — inhalation of xenon in a sub-narcotic dosage
  Arms: Main group
Other: premedication hydroxyzine 25 mg — taking anxiolytic 30 minutes before surgery
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to propose for implementation and evaluate the effectiveness of xenon sedation for the relief of psychoemotional stress disorder before the operation of refractive laser vision correction patients with high anxiety and stress instability who underwent xenon analgosedation before refractive laser vision correction. The main question[s] it aims to answer are:

1. To develop a method of xenon sedation in patients with a high level of psychoemotional stress before surgery - refractive laser vision correction.
2. To evaluate the effect of inhaled xenon anesthesia in a sub-narcotic dose on the duration of surgery, satisfaction of surgeons and patients with anesthesia, the level of postoperative pain in patients in comparison with anxiolytics.

The following will be studied: the level of preoperative anxiety, the dynamics of glycemia and blood cortisol levels, heart rate variability, electrical microamplitudes of the ECG signal, the anti-stress and analgesic effect of xenon.

If there is a comparison group: the researchers will compare [the group with xenon sedation and the control group] to see if there is [an anti-stress effect of xenon in patients before laser vision correction].

DETAILED DESCRIPTION:
The aim of the study is to propose for implementation and evaluate the effectiveness of xenon sedation for the relief of psychoemotional stress disorder before the operation of refractive laser vision correction.

Research objectives

1. To develop a method of xenon sedation in patients with a high level of psychoemotional stress before surgery - refractive laser vision correction.
2. To evaluate the effect of inhaled xenon anesthesia in a sub-narcotic dose on the duration of surgery, satisfaction of surgeons and patients with anesthesia, the level of postoperative pain in patients in comparison with anxiolytics.
3. To study the dynamics of laboratory stress markers during xenon sedation before refractive laser vision correction operations, in comparison with anxiolytics of the non-benzodiazepine series.
4. To evaluate the change in heart rate variability indicators on the "Varicard" devices and the "Cardiovisor" software package (ECG dispersion mapping method) in comparison with the anxiolytics of the non-benzodiazepine series in the studied groups of patients.
5. To study the economic component in the expenditure of an inhalation anesthetic during xenon anesthesia in a sub-narcotic dosage in outpatient ophthalmic surgery.

The studied phenomena are: the level of preoperative anxiety, the dynamics of glycemia and blood cortisol levels, heart rate variability, electrical microamplitudes of the ECG signal, the anti-stress and analgesic effect of xenon.

The object of the study:

The main group (patients with high anxiety and stress instability, who underwent xenon analgosedation before refractive laser vision correction) - 70 people.

The control group (patients with high anxiety and stress instability, who underwent local anesthesia using standard premedication with hydroxyzine (hydroxyzine) 25 mg.) - 70 people.

Inclusion criteria:

* upcoming surgery in the form of laser vision correction (Femto Lasik or ReLEx ® SMILE);
* male and female patients over 18 years of age with high anxiety and stress instability (Spielberger-Khanin test of 46 points or more);
* signed informed consent to participate in the study.

Non-inclusion criteria:

• concomitant somatic diseases in the decompensation stage.

Exclusion criteria:

• the patient's desire to withdraw from the study;

Research methods:

1. Assessment of stress levels by testing on the Spielberger-Hanin scale.
2. Examination of the patient on a Cardiovisor and Varicard before and after surgery.
3. Laboratory assessment of the level of capillary glucose and cortisol in the blood before and after surgery.
4. Assessment of postoperative pain on a visual-analog scale.
5. Statistical methods. Practical significance: the use of xenon sedation to relieve the psychoemotional tension of patients during the operation ReLEx® SMILE and Femto Lasik will reduce the frequency of complications of these operations (loss of vacuum fixation). The proposed method will also expand the availability of such operations for patients with increased neuro-reflex excitability.

Novelty of the study:

In this study, for the first time, there will be:

1. The method of application of xenon sedation for relief of psychoemotional tension of patients during operations - refractive laser vision correction (ReLEx® SMILE and Femto Lasik) will be presented.
2. The method of assessing the autonomic nervous system (Varicard) will be used for the first time to control the dynamics of stress in ophthalmic surgery using xenon sedation.
3. The method reflecting changes in the electrophysiological state of the myocardium (Cardiovisor) under the influence of xenon sedation will be used for the first time.

ELIGIBILITY:
Inclusion Criteria:

* upcoming operation ReLEx® SMILE;
* high anxiety and stress instability (Spielberger-Khanin test of 46 points or more);
* signed informed consent to participate in the study.

Exclusion Criteria:

- concomitant somatic diseases in the decompensation stage.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
the concentration of cortisol in the blood | 30 minutes before surgery and 30 minutes after surgery
  the change in the cortisol concentration index as a stress marker during xenon sedation before refractive laser vision correction operations in comparison with anxiolytics of the non-benzodiazepine series.
glucose concentration in capillary blood | 30 minutes before surgery and 30 minutes after surgery
  changes in glucose concentration index as a stress marker during xenon sedation before refractive laser vision correction operations in comparison with anxiolytics of the non-benzodiazepine series.
stress index | 30 minutes before surgery and 30 minutes after surgery
  the change in the heart rate variability measured by the Varikard device in comparison with the anxiolytics of the non-benzodiazepine series in the studied groups of patients.
rhythm index | 30 minutes before surgery and 30 minutes after surgery
  the change in the rhythm index measured by the Cardiovisor device in comparison with benzodiazepine-type anxiolytics in the studied groups of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Sergey Sakhnov, Study Director — Director
Locations (1):
- s. Fyodorov Eye Microsurgery Federal State Inctitution, Krasnodar, Russia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Duygu Yalinbas, Erman Bozali, Ayla Uzun Çiçek. Comparison of Self-Esteem and Social Anxiety Levels of Adolescents Who Wear Spectacles and Who Do Not. Turkish Journal of Family Medicine & Primary Care.2021; 15(4):862-871. https://doi.org/10.21763/tjfmpc.976914
- [Background] Nazari R, Ahmadzadeh R, Mohammadi S, Rafiei Kiasari J. Effects of hand massage on anxiety in patients undergoing ophthalmology surgery using local anesthesia. J Caring Sci. 2012 Aug 25;1(3):129-34. doi: 10.5681/jcs.2012.019. eCollection 2012 Sep. PMID 25276687
- [Background] Hou H, Li X, Song Y, Ji Y, Sun M, Wang D, Jiao J, Qu J, Gu H. Effect of interactive, multimedia-based home-initiated education on preoperative anxiety inchildren and their parents: a single-center randomized controlled trial. BMC Anesthesiol. 2023 Mar 28;23(1):95. doi: 10.1186/s12871-023-02055-7. PMID 36977985
- [Background] Hatam Boustani, Sirus Pakseresht, Mitra Zamani, Mohammad Akmali. The effect of music therapy on the anxiety level of patients undergoing LASIK eye surgery before operation. Minerva Medica. 2018. 5(7): 80-87. https://doi.org/10.23736/S0394-9508.17.04756-8
- [Background] Sasajima H, Zako M, Ueta Y, Murotani K. Effects of Low-Concentration Nitrous Oxide Anesthesia on Patient Anxiety During Cataract Surgery: A Retrospective Cohort Study. Clin Ophthalmol. 2022 Aug 24;16:2803-2812. doi: 10.2147/OPTH.S382476. eCollection 2022. PMID 36042911
- [Background] Shah R. History and Results; Indications and Contraindications of SMILE Compared With LASIK. Asia Pac J Ophthalmol (Phila). 2019 Sep-Oct;8(5):371-376. doi: 10.1097/01.APO.0000580132.98159.fa. PMID 31567264
- [Background] Ganesh S, Brar S, Arra RR. Refractive lenticule extraction small incision lenticule extraction: A new refractive surgery paradigm. Indian J Ophthalmol. 2018 Jan;66(1):10-19. doi: 10.4103/ijo.IJO_761_17. PMID 29283117
- [Background] Xia Y, Fang H, Xu J, Jia C, Tao G, Yu B. Clinical efficacy of xenon versus propofol: A systematic review and meta-analysis. Medicine (Baltimore). 2018 May;97(20):e10758. doi: 10.1097/MD.0000000000010758. PMID 29768360